CLINICAL TRIAL: NCT02070692
Title: Tamoxifen for the Treatment of Unfavorable Bleeding Patterns in Etonogestrel Contraceptive Implant Users
Brief Title: Tamoxifen for the Treatment of Unfavorable Bleeding in Contraceptive Implant Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Katharine Simmons, MD, Fellow in Family Planning, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SFPRF14-1; SFPRF14-1 (Other Grant/Funding Number: Society of Family Planning)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Menstruation Disturbances
Keywords: Contraceptive implant; Irregular vaginal bleeding; Etonogestrel implant
MeSH Terms: conditions — Menstruation Disturbances | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamoxifen (Experimental): Participants will be randomized to receive either tamoxifen 10mg twice daily for seven days, or placebo twice daily for seven days, to be started on the third day of an episode of bleeding.
  Interventions: Drug: Tamoxifen
- Placebo (Placebo Comparator): Placebo tablets twice daily for seven days, to be started on the third day of a bleeding episode.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamoxifen — 7 day course of tamoxifen during an episode of irregular vaginal bleeding
  Other Names: Nolvadex
  Arms: Tamoxifen
Drug: Placebo — 7 day course of placebo during an episode of irregular vaginal bleeding
  Arms: Placebo

SUMMARY:
The purpose of this study is to study whether a drug called tamoxifen can reduce vaginal bleeding in women who are using the Etonogestrel contraceptive implant.

DETAILED DESCRIPTION:
Nearly all of the 3 million unintended pregnancies in the United States each year result from inconsistent or non-use of contraception. Increasing use of the most effective methods of contraception will reduce unintended pregnancies and their social, medical and economic consequences. The contraceptive etonogestrel implant (ENG implant) is 20 times more effective at pregnancy prevention than oral contraceptive pills, but it has bleeding side effects that make it unappealing for many women. Tamoxifen, a selective estrogen receptor modulator (SERM) used most commonly for adjuvant treatment of breast cancer, has previously been shown to dramatically reduce bleeding in users of an older levonorgestrel-based contraceptive implant (Norplant tm). It has not been studied in newer progestin-based methods such as the ENG implant. If tamoxifen could stop bleeding in users of the ENG implant, it would give patients and physicians a valuable option for management of progestin-induced irregular bleeding. This research project will test the effectiveness of tamoxifen taken on an as-needed basis to treat abnormal bleeding in ENG implant users. If tamoxifen can be established as an effective treatment for frequent or prolonged bleeding, it will increase the acceptability of the ENG implant, increase its use and reduce unintended pregnancies. This is the first project to evaluate tamoxifen for treatment of unfavorable bleeding in users of the ENG contraceptive implant.

ELIGIBILITY:
Inclusion Criteria:

* Current user of the etonogestrel implant (Nexplanon, Implanon) for at least one month
* Experiencing bleeding episodes more frequently than every 24 days, or a single episode of bleeding lasting longer than 14 days
* English or Spanish speaking
* Planning to continue implant use for six months
* Access to a cell phone that can accept and send text messages

Exclusion Criteria:

* Postpartum within six months
* Post-abortion within six weeks
* Pregnant
* Breast-feeding
* Undiagnosed abnormal uterine bleeding pre-dating placement of contraceptive implant
* Bleeding dyscrasia
* Anticoagulation use
* Active cervicitis
* Allergy to tamoxifen
* History of venous thromboembolism
* Current or past breast or uterine malignancy
* Use of medication contraindicated with tamoxifen (coumadin, letrozole, bromocriptine, rifampicin, aminoglutethimide, phenobarbital)

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study under review for publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamoxifen | Placebo
Started | 28 | 28
Completed | 18 | 16
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Full Range); unit: years] | 25.4 [18 to 36] | 23.9 [15 to 38] | 24.6 [15 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 3 | 4
  White | 25 | 20 | 45
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 2
Days of bleeding/spotting in 30 days prior to enrollment [Mean (Standard Deviation); unit: days] | 17.3 (8.5) | 22.2 (6.6) | 19.75 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Days
Description: The primary objective of this study is to determine whether tamoxifen taken by users of the ENG implant on an as-needed basis for frequent or prolonged bleeding can reduce the number of bleeding days by at least 40% over 180 days, when compared to placebo.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 18 | 16
days | 65.6 (37.5) | 46.9 (28.1)

2. Primary Outcome: Bleeding/Spotting Days
Description: Bleeding/spotting days
Time Frame: 30 days
Population: Number of patients analyzed is number of patients who completed 30 days of follow up. Two subjects in the tamoxifen arm and three in the placebo arm were lost to follow up prior to 30 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 26 | 25
days | 10.5 (9.0) | 15.5 (8.5)

3. Primary Outcome: Consecutive Bleeding-free Days After Study Drug
Description: Consecutive bleeding-free days after study drug
Time Frame: up to 180 days
Population: Number of subjects analyzed is the number of subjects who started taking the study drug. One subject in the tamoxifen arm and there in the placebo arm did not initiate study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 27 | 25
days | 28.8 (24.5) | 13.6 (19.2)

4. Secondary Outcome: Satisfaction (as Recorded on a 100mm Visual Analog Scale Where 0 is Not at All Satisfied and 100mm is Completely Satisfied)
Description: Secondary objective is to determine whether tamoxifen can improve satisfaction with the implant and with bleeding patterns.
Time Frame: 180 days
Population: Number of subjects analyzed is the number of subjects who completed a final study visit (either completion of full study or early termination visit) to provide a final estimation of satisfaction.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 22 | 21
units on a scale | 61.4 (24.7) | 53.6 (33.3)

5. Secondary Outcome: Number of Participants Experiencing Ovulation After First Use of Study Drug
Description: A third secondary objective is to determine whether taking tamoxifen at this dose compromises ovulation suppression in ENG users. Tamoxifen is known to transiently raise serum estradiol levels, but does not affect gonadotropin release in premenopausal women. Therefore, it is unlikely to interact with the ovulation suppression provided by the implant. However, to further investigate any theoretical interaction between tamoxifen and etonogestrel, urine markers of ovulation will be collected to document ongoing ovulation suppression with intermittent tamoxifen use.
Time Frame: 30 days
Population: Number of subjects analyzed are those that provided urine samples. No subject who provided urine samples was excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Tamoxifen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No